CLINICAL TRIAL: NCT02394483
Title: F901318 - A Phase I, Double-Blind, Placebo Controlled, Single Ascending Oral Dose, Safety, Tolerability and Pharmacokinetic Study in Healthy Male Subjects
Brief Title: Single Ascending Oral Dose Study of F901318
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: F2G Biotech GmbH (Industry)
Collaborators: Simbec-Orion Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F901318-01-03-15
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-08

CONDITIONS: Invasive Aspergillosis
Keywords: Single ascending dose; double blind
MeSH Terms: interventions — Metabolism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- Cohort A active (Experimental): 2 mg/kg orally F901318 safety,F901318 tolerability and F901318 pharmacokinetics
  Interventions: Drug: F901318 safety; Drug: F901318 tolerability; Drug: F901318 pharmacokinetics
- Cohort A placebo (Placebo Comparator): Matching placebo safety,placebo tolerability and placebo pharmacokinetics
  Interventions: Other: Placebo safety; Other: Placebo tolerability; Other: Placebo pharmacokinetics
- Cohort B active (Experimental): 4 mg/kg orally F901318 safety,F901318 tolerability and F901318 pharmacokinetics
  Interventions: Drug: F901318 safety; Drug: F901318 tolerability; Drug: F901318 pharmacokinetics
- Cohort B placebo (Placebo Comparator): Matching placebo safety,placebo tolerability and placebo pharmacokinetics
  Interventions: Other: Placebo safety; Other: Placebo tolerability; Other: Placebo pharmacokinetics
- Cohort C active (Experimental): 6 mg/kg orally F901318 safety,F901318 tolerability and F901318 pharmacokinetics
  Interventions: Drug: F901318 safety; Drug: F901318 tolerability; Drug: F901318 pharmacokinetics
- Cohort C placebo (Placebo Comparator): Matching placebo safety,placebo tolerability and placebo pharmacokinetics
  Interventions: Other: Placebo safety; Other: Placebo tolerability; Other: Placebo pharmacokinetics
- Cohort D active (Experimental): 8 mg/kg orally F901318 safety,F901318 tolerability and F901318 pharmacokinetics
  Interventions: Drug: F901318 safety; Drug: F901318 tolerability; Drug: F901318 pharmacokinetics
- Cohort D placebo (Placebo Comparator): Matching placebo safety,placebo tolerability and placebo pharmacokinetics
  Interventions: Other: Placebo safety; Other: Placebo tolerability; Other: Placebo pharmacokinetics
- Cohort E active (Experimental): 10 mg/kg orally F901318 safety,F901318 tolerability and F901318 pharmacokinetics
  Interventions: Drug: F901318 safety; Drug: F901318 tolerability; Drug: F901318 pharmacokinetics
- Cohort E placebo (Placebo Comparator): Matching placebo safety,placebo tolerability and placebo pharmacokinetics
  Interventions: Other: Placebo safety; Other: Placebo tolerability; Other: Placebo pharmacokinetics

INTERVENTIONS:
Drug: F901318 safety — Safety assessments
  Other Names: adverse events
  Arms: Cohort A active; Cohort B active; Cohort C active; Cohort D active; Cohort E active
Drug: F901318 tolerability — Tolerability assessments
  Other Names: adverse events
  Arms: Cohort A active; Cohort B active; Cohort C active; Cohort D active; Cohort E active
Drug: F901318 pharmacokinetics — Pharmacokinetic assessments
  Other Names: metabolism
  Arms: Cohort A active; Cohort B active; Cohort C active; Cohort D active; Cohort E active
Other: Placebo safety — Safety assessments
  Other Names: adverse events
  Arms: Cohort A placebo; Cohort B placebo; Cohort C placebo; Cohort D placebo; Cohort E placebo
Other: Placebo tolerability — Placebo tolerability
  Other Names: adverse events
  Arms: Cohort A placebo; Cohort B placebo; Cohort C placebo; Cohort D placebo; Cohort E placebo
Other: Placebo pharmacokinetics — Plaacebo pharmacokinetics
  Other Names: metabolism
  Arms: Cohort A placebo; Cohort B placebo; Cohort C placebo; Cohort D placebo; Cohort E placebo

SUMMARY:
Double blind, placebo controlled, ascending single oral dose, sequential group study. Forty subjects will complete the study in 5 cohorts (Groups A to E), each group consisting of 8 subjects. Each subject will be on study for approximately 6 weeks. Each subject will participate in one treatment cohort only, residing at the Clinical Research Unit (CRU) from Day -1 (the day before dosing) to Day 6 (120 hours post-dose). Each cohort will be dosed in a leading edge design in which two subjects will receive study drug (1 active and 1 placebo) on the first dosing day, and the last 6 will receive study drug (5 active and 1 placebo) on the second dosing day.

All subjects will return for a post-study visit 8 to 10 days after the dose of study medication.

Cohorts will be dosed at 2 weekly intervals. There will be a review of safety data, after the first two subjects have been dosed and before dosing of the subsequent six subjects. There will be a complete review of safety and pharmacokinetic data of each cohort prior to each dose escalation.

DETAILED DESCRIPTION:
Male healthy subjects conforming to the selection criteria will be invited to take part in the study.

Screening visit (Visit 1) After giving fully informed, written consent, subjects will attend the clinic.

Subjects will undergo screening within 28 days prior to the first dose administration. Prior to the screening visit, subjects will:

* Refrain from vigorous exercise for 7 days
* Abstain from alcohol for 48 hours
* Subjects will sign the consent form in the presence of a CRU physician prior to any screening procedures being performed. The information recorded for all subjects, regardless of their suitability for the study, will be retained and archived

The following information and procedures will be recorded and performed as part of the screening assessments:

* Medical history
* Ethnic origin, sex, age, height, weight, and BMI
* Vital signs: supine blood pressure, supine pulse rate, and oral body temperature
* Resting 12 lead ECG
* Physical examination
* Urine drugs of abuse screen, cotinine and breath alcohol
* Fasting clinical laboratory and serology investigations

Up to 28 days after screening, subjects will attend the clinic. Subjects will be admitted to the research unit at approximately 13:00 hours in the afternoon the day before dosing (Day -1; -19 hours pre-dose). Urine will be subjected to a screen for drugs of abuse and there will be a breath test for alcohol and cotinine. Detection of any of these substances will disqualify the subject from the study. A physical examination, check of inclusion/exclusion criteria, clinical laboratory evaluations, oral temperature and body weight will be performed. Subjects will be asked whether they have experienced any adverse events or taken any concomitant medication since their previous visit. Supper will be served starting at 19.30 hours and a snack at 21.00 hours, following which subjects will be fasting. Water will be allowed ad libitum throughout.

On day 1, the total first urine void of the morning for each subject will be collected into a polyethylene container and, from this, a sample will be taken for urinalysis and pre-dose / baseline F901318 concentration. Within one hour before dosing commences (-1 hour), blood will be drawn for laboratory safety assessments (haematology and clinical chemistry), and pre-dose baseline F901318 and metabolites concentration. Supine and standing blood pressure and pulse rate in triplicate, body temperature and a 12-lead ECG will be recorded. The subjects will also be connected to continuous ECG recording from -1 hour until 12 hours after the start of dosing.

Subjects will be asked whether they have experienced any adverse events overnight. Any concomitant medications will be recorded.

Option 1: Subjects will then be dosed. This will be oral ingestion of a liquid formulation followed by 250 mL of water. Subjects will be dosed with regular (at least 5 minute) intervals between each subject.

After initial dosing, the following measurements and observations will be obtained:

• Blood samples for analysis of F901318 plasma concentration will be drawn at 15, 30, 45, 60, 75, 90, 120 minutes, then 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96 and 120 hours following dosing. Pharmacokinetic blood samples will be analysed and reviewed before each dose escalation. After the first dose administration, the timing of each blood sample may if necessary be adjusted within the 120-hour period for the subsequent dose escalation. The basis for this decision will depend upon the pharmacokinetic profiles obtained from the preceding group of subjects. All changes will be documented in a file note. The number of samples or volume of blood drawn must not be increased without prior approval of the relevant ethics committee.

Option 2: If it appears from pharmacokinetic measurements that oral absorption is extremely rapid, leading to a high Cmax with a relatively low AUC0-12, the dose may be split in half, with the second half being given 4-8 hours after the first. Under these circumstances, the blood sampling schedule would be decided prior to dosing but would not exceed 26 samples over a 120 hour period.

For Both Options:

* Blood samples for analysis of metabolites will be drawn 4 and 8 hours after initial dosing.
* Blood will be collected for safety measurements (haematology and clinical chemistry) 24, 48 and 72 hours post initial dosing.
* Complete urine collections for analysis of F901318 urine concentration will be made for the following intervals in relation to dosing: 0-4, 4-8, 8-12, 12-16, 16-24, 24-48, 48-72, 72-96 and 96-120 hours after initial dosing.
* Supine and standing pulse rate and blood pressure; and body temperature (vital signs) will be recorded 30, 60 and 120 minutes, 4, 8, 24, 48 and 72 hours after initial dosing.
* Twelve-lead ECGs will be obtained 1, 4, 24, 48 and 72 hours after initial dosing.
* The continuous ECG recording will cease 12 hours after initial dosing.
* Spontaneously reported adverse events will be noted throughout.
* A urine sample will be taken for urinalysis 24, 48 hours and 72 hours after initial dosing.
* Lunch will be served approximately 4 hours after initial dosing but after all the 4 hour observations and blood sampling have been completed and a main meal will be served approximately 8 hours and a snack approximately 12 hours after dosing.

Subjects may leave the Research Unit on Day 6, unless they have experienced adverse events that, in the opinion of the Investigator, warrant further observation and/or treatment.

All subjects will be followed up 8-10 days after dosing with a post-study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be males of any ethnic origin between 18 and 45 years of age and with a body weight of 60-100 kg inclusive.
2. Subjects must be in good health, as determined by a medical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations (congenital non haemolytic hyperbilirubinaemia is acceptable).
3. Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions.

Exclusion Criteria:

1. Male subjects who are not willing to use appropriate contraception (such as a condom) during the study and until follow up.
2. Subjects who have received any prescribed systemic or topical medication within 14 days of the dose administration unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety.
3. Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days of the dose administration (with the exception of vitamin/mineral supplements) unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety.
4. Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of the dose administration unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety.
5. Subjects who are still participating in a clinical study (e.g. attending follow-up visits) or who have participated in a clinical study involving administration of an investigational drug (new chemical or biological entity) in the past 3 months.
6. Subjects who have donated any blood, plasma or platelets in the 2 months prior to screening or who have made donations on more than two occasions within the 12 months preceding the dose administration.
7. Subjects with a significant history of drug allergy as determined by the Investigator.
8. Subjects who have any clinically significant allergic disease (excluding non-active hay fever) as determined by the Investigator.
9. Subjects who have a supine blood pressure and supine pulse rate higher than 140/90 mmHg and 100 beats per minute (bpm), respectively, or lower than 90/50 mmHg and 40 bpm, respectively, confirmed by a repeat assessment.
10. Subjects who consume more than 28 units of alcohol per week or who have a significant history of alcoholism or drug/chemical abuse as determined by the Investigator (one unit of alcohol equals ½ pint [285 mL] of beer or lager, one glass [125 mL] of wine, or 1/6 gill [25 mL] of spirits).
11. Subjects with a positive urine drug screen or alcohol breath test result at screening or first admission.
12. Subjects must not have smoked for 3 months prior to first dose administration unless otherwise specified by the Investigator or Sponsor.
13. Subjects with, or with a history of, any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, ocular (including minor trauma) haematological or other major disorders as determined by the Investigator.
14. Subjects who are known to have serum hepatitis, or who are carriers of the hepatitis B surface antigen (HBsAg) or hepatitis C antibody, or who have a positive result to the test for HIV antibodies.
15. Subjects who have an abnormality in the 12-lead ECG that, in the opinion of the Investigator, increases the risk of participating in the study, such as QTcB interval >430 msec, 2nd or 3rd degree atrioventricular block, complete left bundle branch block, complete right bundle branch block or Wolff-Parkinson-White Syndrome, defined as PR<110 msec, confirmed by a repeat ECG.
16. Subjects who, in the opinion of the Investigator, should not participate in the study for any other reason.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Safety (Adverse events) | 10 days
  Adverse events

SECONDARY OUTCOMES:
Tolerability (Adverse events) | 10 days
  Adverse events
Pharmacokinetics (Area under concentration time curve, AUC) | 120 hours
  Area under concentration time curve
Pharmacokinetics (Cmax) | 12 hours
  Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Girish Sharma, Principal Investigator — Simbec Orion Ltd
Locations (1):
- Simbec Orion, Merthyr Tydfil, Wales, United Kingdom